CLINICAL TRIAL: NCT05424224
Title: Using Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Depression
Brief Title: Using rTMS to Treat Depression
Status: Active, not recruiting | Type: Observational
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Malek Adjouadi, PhD, Professor, Florida International University
Other Study IDs: IRB-18-0298-CR03
Record Dates: First submitted 2022-05-17; First posted 2022-06-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: Depression; rTMS; EEG
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- patients with depression: patients with depression
  Interventions: Device: MagVita

INTERVENTIONS:
Device: MagVita — rTMS system

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a promising, novel, non-invasive therapy for depression. In fact, there is an FDA-approved depression protocol to stimulate the dorsolateral prefrontal cortex (dlPFC). Its efficacy and safety have improved significantly with continued research and clinical experience. However, it is not known how to identify potential patients who would benefit most from treatment.

The primary goal of this study is to determine if changes in specific electroencephalogram (EEG) parameters after treatment can predict whether patients are responders or non-responders to rTMS. The second objective is to analyze changes in the functional connectivity of specific brain regions in responders compared to non-responders.

The hypothesis is that through rTMS treatment, investigators will be able to increase the activity in the frontal region that includes the dorsolateral prefrontal cortex (DLPFC). Scalp EEG signals will be processed in order to compare EEG brain connectivity and Frontal alpha asymmetry index (FAA) to determine if there are differences before and after the treatment. EEG FAA is usually calculated by subtracting the right-side EEG power estimates from the respective counterpart on the other side. According to literature, depressive patients seem to have comparatively higher left frontal alpha power. Cortical activity is related to a reduced EEG power, which is reflected in depressed subjects. On the other hand, higher alpha power could also be interpreted as inhibition.

Investigators will try to delineate changes in resting EEG functional connectivity before and after high-frequency left prefrontal rTMS, by using biomarkers such as: time/frequency connectivity, Alpha asymmetry index, among others. TMS also allows cortical properties, such as excitability, inhibition, oscillatory activity and connectivity to be directly probed within a specific region of the cortex. Other studies suggest that alterations in gamma oscillations in the dorsolateral prefrontal cortex and neighboring frontal regions are also potential shared biomarkers in psychiatry, highlighting the potential of EEG signals to help identify suitable biomarkers. Given its relative low cost and ease of use, when compared to brain imaging tools such as magnetic resonance imaging (MRI) or positron emission tomography (PET), EEG could be added to the clinical study so that precise neurophysiological changes before and after treatments can be assessed.

DETAILED DESCRIPTION:
rTMS treatment for subjects who are suffering depression and are suitable for rTMS according to the inclusion and exclusion criteria using the FDA MagVenture: MagVita TMS system. This protocol will be conducted following the safety guidelines in order to minimize risk. Dr. Patricia Junquera will be present during the TMS sessions.

For this research study investigators are recruiting patients with depression. Two groups will be created:

Group 1 = Research-onlyGroup; with 2 sub-group: 1-A= TMS treatment up to 6 weeks and 1-B = SHAM 2 weeks + TMS treatment up to 4 weeks.

Group 2 = Treatment + research group, If voluntarily consenting, patients who obtain clinical treatment for depression with TMS at FIU Ambulatory Care Center (ACC) will have EEG, recorded (duration: 20min).

Group 1= Sub-Group 1-A and Sub-Group 1-B Sub-Group 1-A = Research intervention: ten patients will receive active rTMS during 6 weeks (30 sessions). EEG will be recorded before rTMS sessions during session 1, 10, and 30.

Sub-Group 1-B= Sham and research intervention : Blind-randomized trial 10 sessions of sham-controlled rTMS will be apply to ten patients, after the 2 weeks group 1-B would be incorporated for 4 weeks to the same protocol that group 1-A (Activer TMS). EEG will be acquire before the first session and after session 10 to compare and evaluate the efficacy of rTMS in depression for these two groups during the first two weeks.

Group 2 = Clinical Treatment + research group: If voluntarily consenting, patients who obtain clinical treatment for depression with TMS at FIU Ambulatory Care Center (ACC) will have EEG recorded at the beginning of treatment, session 10, session 20, and at the end of the protocol, session 30 (duration: 19 min).

Motor Threshold (MT) Determination has two purposes: to determine the location of the hand area of the motor cortex and to determine stimulation level. Once the motor cortex is found, a line is drawn on the patient's individual cap to show the operator where to place the coil when performing the actual depression treatments. The MT determination is performed on the left hemisphere because the subsequent depression treatments are performed over the left dorsolateral prefrontal cortex (DLPFC). When performing rTMS depression treatment, the stimulation level is defined as 120 % of MT

Treatments Steps:

Initial session with Motor Threshold (MT) determination, followed by 5 treatment sessions per week during a period of normally 2-6 weeks.

EEG recordings will be performed using the Xltek EEG (Electroencephalograph) system, designed for quick and convenient hook-up, it will record the brain's spontaneous electrical activity and evoked responses non-invasively from the scalp. Approximately 10-20 minutes of resting-state EEG will be recorded before rTMS sessions during session 1, 10 and 30).

Study will be conducted at ACC 145-145-A clinical facility, During treatment sessions, the patient is comfortably seated in the treatment chair with a vacuum pillow around the neck to provide optimal support of the head.

The study is of minimal risk with occasional side effects of the test are minor and brief headache from prolonged TMS stimulation.

Response and Treatment Protocol in case of Seizure:

In case a patient suffers the occurrence of a seizure during an rTMS session, the following steps are undertaken:

•If a seizure occurs, testing (TMS) will be postponed at least 1 hour, or until baseline function returns.

The significance of this work is to create a new understanding of the therapeutic effect of rTMS in participants with depression, using EEG to assess the lasting effects of the treatment. This can lead us to the creation of a maintenance protocol to prolong the effects of rTMS in this population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Depression
* must be willing to cooperate.

Exclusion Criteria:

* implanted electronic devices (e.g., pacemaker, medication pump, brain or vagus nerve stimulator, cochlear implant)
* history of seizures
* intracranial metal (e.g., aneurysm clip)
* inability of the participant to cooperate with the Transcranial Magnetic Stimulation (TMS) session

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult with symptoms of depression.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
EEG parameters to asses the change | Session 1(baseline), Session 10 ( after 2 weeks of treatment), and 30 ( treatment completion)
  Resting-state Electroencephalogram (EEG) can serve as an assessment signal that will determine the benefits of the treatment and the efficacy of this procedure. Frequency domain features will be extracted to analyze the change over the time of the treatment. Connectivity maps will be derived for the most important frequency bands( Delta, Theta, Alpha, and Beta).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified EEG will be shared to other researches .

REFERENCES:
- [Result] Chu HT, Cheng CM, Liang CS, Chang WH, Juan CH, Huang YZ, Jeng JS, Bai YM, Tsai SJ, Chen MH, Li CT. Efficacy and tolerability of theta-burst stimulation for major depression: A systematic review and meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Mar 2;106:110168. doi: 10.1016/j.pnpbp.2020.110168. Epub 2020 Nov 7. PMID 33166668
- [Result] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Result] Noda Y, Zomorrodi R, Saeki T, Rajji TK, Blumberger DM, Daskalakis ZJ, Nakamura M. Resting-state EEG gamma power and theta-gamma coupling enhancement following high-frequency left dorsolateral prefrontal rTMS in patients with depression. Clin Neurophysiol. 2017 Mar;128(3):424-432. doi: 10.1016/j.clinph.2016.12.023. Epub 2017 Jan 9. PMID 28160748
- [Result] Kelly MS, Oliveira-Maia AJ, Bernstein M, Stern AP, Press DZ, Pascual-Leone A, Boes AD. Initial Response to Transcranial Magnetic Stimulation Treatment for Depression Predicts Subsequent Response. J Neuropsychiatry Clin Neurosci. 2017 Spring;29(2):179-182. doi: 10.1176/appi.neuropsych.16100181. Epub 2016 Nov 30. PMID 27899052